CLINICAL TRIAL: NCT05647265
Title: Official Title Neoadjuvant Immunotherapy in Sarcomatoid Mesothelioma
Brief Title: Testing the Addition of Immunotherapy Before Surgery for Patients With Sarcomatoid Mesothelioma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A082101; NCI-2022-09320 (Other: NCI); U10CA180821 (NIH)
Record Dates: First submitted 2022-11-29; First posted 2022-12-12 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Pleural Biphasic Mesothelioma; Pleural Sarcomatoid Mesothelioma
MeSH Terms: interventions — Nivolumab; Ipilimumab; CTLA-4 Antigen; Surgical Procedures, Operative; Magnetic Resonance Spectroscopy; X-Rays; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (nivolumab, ipilimumab, surgery) (Experimental): Patients receive nivolumab IV, ipilimumab IV, and may undergo surgery on study. Patients also undergo CT or MRI and PET throughout the trial.
  Interventions: Biological: Nivolumab; Biological: Ipilimumab; Procedure: Surgical Procedure; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Biological: Nivolumab — Given IV
  Other Names: 946414-94-4, BMS-936558, CMAB819, MDX-1106, NIVO, NIVOLUMAB, Nivolumab, Nivolumab Biosimilar CMAB819, ONO-4538, Opdivo
Biological: Ipilimumab — Given IV
  Other Names: 477202-00-9, Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody, BMS-734016, IPILIMUMAB, ipilimumab, Ipilimumab Biosimilar CS1002, MDX-010, MDX-010, MDX-CTLA4, Yervoy
Procedure: Surgical Procedure — Undergo surgery
Procedure: Computed Tomography — undergo CT
  Other Names: CAT, CAT Scan,
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: MRI
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, PET, Pet Scan

SUMMARY:
This phase II trial evaluates the safety and effectiveness of giving immunotherapy (nivolumab and ipilimumab) before surgery for controlling disease in patients with stage I-IIIa sarcomatoid mesothelioma. Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving immunotherapy before surgery may be more effective at controlling disease in patients with sarcomatoid mesothelioma than giving immunotherapy alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the percentage of patients with potentially resectable non-epithelioid mesothelioma who are able to proceed with surgery after neoadjuvant ipilimumab and nivolumab.

II. To determine the progression-free survival rate at 12 months after the initiation of neoadjuvant ipilimumab and nivolumab.

SECONDARY OBJECTIVES:

I. To determine the rate of intra-operative or post-operative complications following neoadjuvant immunotherapy.

II. Best response per modified pleural Response Evaluation Criteria in Solid Tumors (RECIST).

III. Major pathologic response rate. IV. Time to recurrence after surgery.

EXPLORATORY OBJECTIVES:

I. To evaluate the association between the change in peripheral T cell clonality relative to baseline and treatment response.

II. To evaluate the association between PD-L1 expression at baseline and treatment response.

III. To evaluate whether a novel mesothelioma immune signature identified by Dr. Mansfield's laboratory is predictive of response.

OUTLINE:

Patients receive nivolumab intravenously (IV), ipilimumab IV, and may undergo surgery on study. Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI) and positron emission tomography (PET) throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Sarcomatoid or sarcomatoid-dominant (> 50%) biphasic, pleural mesothelioma
* Stage: I-IIIA disease per Union for International Cancer Control (UICC) TNM Classification of Malignant Tumours 8th edition
* Measurable disease or non-measurable disease as defined
* No prior treatment which would be considered treatment for the primary neoplasm or impact the primary endpoint
* No treatment with hormones or other chemotherapeutic agents except for hormones administered for non-disease-related conditions (e.g., insulin for diabetes and or hormonal therapy for breast, prostate cancer etc.)
* Not pregnant and not nursing, because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown

  * Therefore, for women of childbearing potential only, a negative pregnancy test done =< 14 days prior to registration is required
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 or Karnofsky >= 60%
* Absolute neutrophil count (ANC) >= 1,000/mm^3
* Leukocytes >= 2,000/mm^3
* Platelet count >= 100,000/mm^3
* Creatinine =< 1.5 x upper limit of normal (ULN) OR creatinine clearance >= 40 mL/min
* Total bilirubin =<1.5 x ULN, except patients with Gilbert Syndrome who can have total bilirubin < 3.0 mg/dl
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3.0 x ULN
* Alkaline (alk) phosphatase (phos) =< 3.0 x ULN
* No active, known or suspected autoimmune disease except for vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
* No active systemic infection requiring therapy, as well as positive tests for hepatitis B surface antigen or hepatitis C antibody
* No history of any other condition that may require the initiation of anti-tumor necrosis factor alpha (TNFalpha) therapies or other immunosuppressant medications during the study
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* STEP 2 ELIGIBILITY CRITERIA: Completion of at least 1 cycle of treatment and not have an unresolved adverse event that would preclude surgery
* STEP 2 ELIGIBILITY CRITERIA: No evidence of progression that would preclude resection
* STEP 2 ELIGIBILITY CRITERIA: ECOG performance status =< 2 or Karnofsky >= 60%
* STEP 2 ELIGIBILITY CRITERIA: Predicted forced expiratory volume in 1 second (FEV1) > 35% and postoperative predicted diffusion capacity of the lung for carbon monoxide (DLCO) > 35%
* STEP 2 ELIGIBILITY CRITERIA: Registration to step 2 no less than 21 days and no more than 90 days after the last dose of neoadjuvant therapy

Exclusion Criteria:

* No patients deemed to be unresectable or poor surgical candidates
* No patients with chest wall invasion, peritoneal spread, contralateral pleural involvement, mediastinal organ involvement, vertebral involvement, or metastases to contralateral intrathoracic lymph nodes, or any supraclavicular nodes
* No patients with a history of symptomatic interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Surgery Rate | immediately after the completion of neoadjuvant immunotherapy and surgery
  The rate of surgery after neoadjuvant immunotherapy among the feasibility analysis population as well as the 80% and 95% exact Clopper-Pearson confidence intervals will be estimated.
Progression free survival (PFS) | At 12 months after initiation of neoadjuvant immunotherapy
  PFS will be determined per modified Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. The rate of PFS at 12 months after the initiation of neoadjuvant immunotherapy among the feasibility and efficacy analysis population as well as the 80% and 95% exact Clopper-Pearson confidence intervals will be estimated.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 5 years
  The type of adverse events, the frequency of each type and its grade will be summarized. The frequency and the percentage of severe adverse events will be presented in bar charts over treatment phase (neoadjuvant immunotherapy, surgery) to describe the change of adverse event or complication severity over time. The rates of the pre-operative or post-operative complications (within 30 days of surgery) will be estimated with its exact 95% confidence interval.
Objective response rate | Up to 5 years
  Will be determined per modified RECIST. Response rate will be reported with 95% exact confidence interval.
Major pathologic response | Up to 5 years
  Defined as =< 10% residual viable tumor in the resected lung and lymph node tissue. Response rates will be reported with 95% exact confidence interval.
Time to recurrence | Time from surgery to disease relapse, progression, or second tumor, whichever occurs first, assessed up to 5 years
  Time to recurrence will be estimated among those patients who receive surgery and will be characterized by estimating cumulative incidence function and conducting cause-specific and subdistribution hazard regression.

OTHER OUTCOMES:
Biomarkers | Up to 5 years
  The association of pre-treatment and on-treatment biomarkers in peripheral blood and in tumor tissues with response and time to recurrence, will be evaluated univariately through Chi-square test or log-rank test and through logistic regression model or Cox regression model with other prognostic factors adjusted.

CONTACTS AND LOCATIONS:
Locations (127):
- United States (127):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - PCR Oncology, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Providence Queen of The Valley, Napa, California
  - Providence Medical Foundation - Santa Rosa, Santa Rosa, California
  - Providence Santa Rosa Memorial Hospital, Santa Rosa, California
  - Beebe Medical Center, Lewes, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Christiana Care - Union Hospital, Elkton, Maryland
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Duke University Medical Center, Durham, North Carolina
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Hood River Memorial Hospital, Hood River, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Skagit Regional Health Cancer Care Center, Mount Vernon, Washington
  - Valley Medical Center, Renton, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Cancer Care Northwest-Valley, Spokane, Washington
  - Cancer Care Northwest-North Spokane, Spokane, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington

IPD SHARING:
Plan to Share IPD: Undecided